CLINICAL TRIAL: NCT01377389
Title: A Phase II Study of Ipilimumab PLUS Androgen Depravation Therapy in Castrate Sensitive Prostate Carcinoma
Brief Title: Ipilimumab + Androgen Depravation Therapy in Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to adverse events
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0378; NCI-2011-01125 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-06-17; First posted 2011-06-21 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Castrate sensitive prostate carcinoma; Metastatic prostate carcinoma; Androgen depravation therapy; ADT; Prostate-specific antigen; PSA; Ipilimumab; Yervoy; BMS-734016; MDX010; Leuprolide; Lupron Depot; Leuprolide Acetate; Goserelin; Zoladex; Degarelix; Firmagon
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ipilimumab; Leuprolide; Goserelin; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ipilimumab + ADT (Experimental): Ipilimumab 10 mg/kg intravenous (IV) Weeks 5, 9, 13, and 17 plus Androgen Depravation Therapy (ADT) of either Leuprolide 7.5 mg intramuscular (IM) , Goserelin 3.6 mg subcutaneous (SQ) or Degarelix 80 mg SQ once a month for 8 months beginning Week 1.
  Interventions: Drug: Ipilimumab; Drug: Leuprolide; Drug: Goserelin; Drug: Degarelix

INTERVENTIONS:
Drug: Ipilimumab — 10 mg/kg by vein over 90 minutes once every 4 weeks, for 4 weeks.
  Other Names: Yervoy; BMS-734016; MDX010
Drug: Leuprolide — 7.5 mg intramuscular once a month for 8 months
  Other Names: Leuprolide Acetate; Lupron Depot
Drug: Goserelin — 3.6 mg subcutaneous once a month for 8 months
  Other Names: Zoladex
Drug: Degarelix — 80 mg subcutaneous once a month for 8 months
  Other Names: Firmagon

SUMMARY:
The goal of this clinical research study is to learn if ipilimumab in combination with either Lupron® (leuprolide), Zoladex® (goserelin), or Firmagon® (degarelix) can affect prostate-specific antigen (PSA) levels in patients with prostate cancer. Researchers also want to learn if these drug combinations affect the body's immune system. The safety of these drug combinations will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Ipilimumab is designed to block the activity of cells that decrease the immune system's ability to fight cancer.

Leuprolide, goserelin, and degarelix are designed to help stop the body from making testosterone (a male sex hormone that prostate cancer cells need to survive), which may slow the growth of cancer cells.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive either leuprolide, goserelin or degarelix . The drug you receive will depend on what the doctor thinks is in your best interest and/or which drug your insurance provider will help to cover. Leuprolide is given through a needle in the muscle. Goserelin and degarelix are given through a needle under the skin in the abdomen. Beginning at Week 1, you will receive the drug 1 time every month or every 3 months for up to 8 months. Your doctor will tell you more about which dosing schedule you will use.

You will also receive ipilimumab by vein over about 90 minutes at Weeks 5, 9, 13, and 17. Your blood pressure will be measured every 30 minutes during the infusion, as well as an hour after you are finished receiving the drug.

Study Visits:

Before each dose of ipilimumab, and every 4 weeks for 6 months after the last dose of ipilimumab, and every 12 weeks after that, the following tests and procedures will be performed:

* You will have a physical exam.
* You will be asked about any other drugs and/or treatments you may be receiving.
* You will be asked about any side effects you may have experienced.
* Your performance status will be recorded.
* Blood (about 3 teaspoons) will be drawn for routine tests and to measure your protein, PSA, and testosterone levels, and to check the function of your pancreas, thyroid, and adrenal glands.
* Urine will be collected for routine tests.
* This blood will also be tested for other hormone levels to check the function of your thyroid and adrenal glands (before each dose of ipilimumab and 4 weeks after the last dose only).

Every 12 weeks, you will have the same imaging scans that you had at screening.

Length of Study:

You may receive the study drugs for up to 8 months. You will remain on study for as long as the disease remains stable. You will be taken off study treatment if you have intolerable side effects or if the disease gets worse.

End-of-Study Treatment/Observation Visit:

Within 14 days after your disease gets worse, the following tests and procedures will be performed:

* You will have a physical exam.
* You will be asked about any drugs and/or treatments you may be receiving.
* You will be asked about any side effects you may have experienced.
* Blood (about 3 teaspoons) will be drawn for routine tests. This blood will also be tested to measure your protein, PSA, and testosterone levels, and to check the function of your pancreas, thyroid, and adrenal glands.
* You will have the same imaging scans that you had at screening.

Long-Term Follow-Up:

A member of the study staff will check up on you about every 6 months after your End-of-Study Treatment/Observation Visit. This will consist of a phone call, an e-mail, or a review of your medical and/or other records. If you are contacted by phone, the call will only last a few minutes.

This is an investigational study. Leuprolide, goserelin, and degarelix are FDA approved and commercially available for the treatment of prostate cancer. Ipilimumab is FDA approved and commercially available for melanoma. Its use to treat prostate cancer is investigational.

Up to 48 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed prostate carcinoma.
2. Evidence of metastatic disease on previous bone scan and/or CT scan and/or MRI.
3. Castrate-sensitive disease. Patients already on ADT are eligible as long as the time from initiation of LHRH analog or antagonist is not greater than 1 month AND the total exposure time to the LHRH analog or antagonist will not exceed 8 months (i.e. the effectiveness of current depot LHRH analog or antagonist does not extend beyond 8 months since its initiation).
4. Patients who have received prior hormonal therapy are allowed to participate as long as they have been off hormone ablation for 1.5 times as long as they were on it: e.g. 1) Patients who have received up to 4 months of hormonal ablation are eligible as long as they have been off hormonal ablation for >/= 6 months; 2) Patients who have received 1 year of hormonal ablation are eligible as long as they have been off hormone ablation for >/= 18 months; 3) Patients who have received up to 2 years of hormonal ablation are eligible as long as they have been off hormonal ablation for >/= 3 years have elapsed since its discontinuation.
5. Eastern Cooperative Oncology Group (ECOG) performance status </= 1
6. Patients must have normal organ and marrow function as defined below: a) white blood cell count (WBC) >/= 3000/uL; b) Absolute neutrophil count (ANC) >/= 1500/uL; c) Platelets >/= 100 x 10^3/uL; d) Hemoglobin >/= 9 g/dL; e) Creatinine </= 2mg/dL; f) ALT </= 2.5 x upper limit of normal (ULN) for patients without liver metastases. For patients with liver metastasis ALT </= 5 x ULN is allowed; g) Bilirubin </= 3 x ULN (except for patients with Gilbert's Syndrome, who must have a total bilirubin </= 3mg/dL)
7. Patients included in the study must be >/= 18 years old
8. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Autoimmune disease: Patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) and autoimmune disorders such as rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus or autoimmune vasculitis [e.g., Wegener's Granulomatosis] are excluded from this study.
2. Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of AEs: e.g. a condition associated with frequent diarrhea or chronic skin conditions, recent surgery or colonic biopsy from which the patient has not recovered, or partial endocrine organ deficiencies.
3. Patients with known brain metastases.
4. Patients with small cell carcinoma of the prostate.
5. History of other malignancies, other than nonmelanoma skin cancer or Ta or T1 (low grade) bladder carcinomas, unless in complete remission and off therapy for that disease for at least 5 years.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, history of congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Known HIV, Hepatitis B, or Hepatitis C.
8. Untreated symptomatic spinal cord compressions.
9. Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to one month prior to or after any dose of ipilimumab).
10. Concomitant therapy with any of the following: IL-2, interferon or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids (used in the management of cancer or non-cancer-related illnesses).
11. Previous participation in another ipilimumab clinical trial or prior treatment with a CD137 agonist or CTLA-4 inhibitor or agonist.
12. History of acute diverticulitis, intra-abdominal abscess, GI obstruction, abdominal carcinomatosis or other known risk factors for bowel perforation.
13. Patients who do not agree to practice appropriate birth control methods while on therapy.
14. Concurrent use of 5-alpha reductase inhibitors (finasteride or dutasteride).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06-17 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana M. Aparicio, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients enrolled at MD Anderson Cancer Center between 2011-2013
Pre-assignment Details: All patients were screened according to inclusion and exclusion criteria as outlined per protocol.
Groups:
- Ipilimumab and Androgen Depravation: Participants with castrate sensitive prostate carcinoma
Period: Overall Study
Arm/Group | Ipilimumab and Androgen Depravation
Started | 30
Completed | 27
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Screen failure | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ipilimumab and Androgen Depravation
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: years] | 63 [45 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Progressed After 7 Months of Being on Treatment
Description: Anti-tumor activity assessed through serial PSA measurements (blood tests) at 7 months on treatment. Progression defined as two consecutive PSA values increasing by at least 20% or more from the lowest PSA value for each patient.
Time Frame: at the end of 7 months on treatment
Population: Out of 27 participants, 24 were evaluable for outcome analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab and Androgen Depravation
Number analyzed (Participants) | 24
Participants
  PSA progression at 7 months | 6
  No PSA progression at 7 months | 18

2. Secondary Outcome: The Number of Clonal Expansion of Cluster of Differentiation 8 (CD8) T-cells
Description: CD8 T-cells are known as cytotoxic T-cells or "killer" T-cells. When the resting CD8 T-cells are activated, the activated CD8 T-cells multiple to fight a specific target so creating a group of specifically activated T-cells. This test measured the minimal number of clonal expansions of CD8 T-cells that always preceded an adverse response to treatment that was due to increased activity in the immune system itself. The minimal number of clonal expansion points to what this increased activity in the immune system might look like.
Time Frame: Each evaluable patient was followed from the time of their first dose until 30 days after their last dose of study drug
Population: 9 were evaluable for outcome analysis out of 11 participants
Measure: Number; unit: clonal expansions
Arm/Group | Ipilimumab and Androgen Depravation
Number analyzed (Participants) | 9
clonal expansions | 55

3. Secondary Outcome: Time to Testosterone Recovery (> 50ng/mL) in Patients Treated With Intermittent ADT Plus Ipilimumab.
Description: The presence of testosterone was followed in each patient from the start of treatment until the testosterone lab test was found to be at a value greater than 50ng/mL.
Time Frame: 1 month up to 7 months.
Population: Out of 27 participants, 24 were evaluable for outcome analysis.
Measure: Mean (Full Range); unit: months
Arm/Group | Ipilimumab and Androgen Depravation
Number analyzed (Participants) | 24
months | 3.4 [1.3 to 6.6]

4. Secondary Outcome: Time to Progression of Disease (PD) Off Androgen Depravation Therapy (ADT), After Treatment With Intermittent ADT Plus Ipilimumab.
Description: The number of months after the last ADT dose until the PSA progression
Time Frame: 2 to 45 months
Measure: Mean (Full Range); unit: months
Arm/Group | Ipilimumab and Androgen Depravation
Number analyzed (Participants) | 18
months | 8.0 [2 to 45.3]

5. Secondary Outcome: The Total Number of Study Drug Related Events Indicated by the Participants
Description: The total number of adverse events which were related to one of the study drugs. Grade 1- Mild, asymptomatic of mild symptoms; clinical or diagnostic observation only; intervention not indicated. Grade 2- Moderate, minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental (daily living activities). Grate 3- Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care of daily life activities.
Time Frame: From the first dose to the last follow-up, up to 60 months
Measure: Number; unit: related events
Arm/Group | Ipilimumab and Androgen Depravation
Number analyzed (Participants) | 27
related events
  Grade 1 | 113
  Grade 2 | 55
  Grade 3 | 25

6. Secondary Outcome: Overall Survival
Description: Overall survival of patients treated with intermittent ADT and ipilimumab in months.
Time Frame: From the date of randomization until the date of first documented progression or date of death from any case, whichever came first, assessed up to 70 months.
Population: Only 22 was analyzed, 5 were uncensored.
Measure: Mean (Full Range); unit: months
Arm/Group | Ipilimumab and Androgen Depravation
Number analyzed (Participants) | 22
months | 36 [14.2 to 53]

ADVERSE EVENTS:
Time Frame: Adverse events collected prior to each dose every 4 weeks for 6 months after the last dose is administered.
Description: Adverse events are documented according to protocol requirements.
Arm/Group | Ipilimumab and Androgen Depravation
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 10/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipilimumab and Androgen Depravation (N=27)
ALT (Hepatobiliary disorders) | 1 (1)
AST (Hepatobiliary disorders) | 1 (1)
Renal Insufficiency (Renal and urinary disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Edema (Vascular disorders) | 1 (1)
CNS Cerebrovascular ischemia (CVA) (Nervous system disorders) | 1 (1)
Adrenal Insufficiency (Renal and urinary disorders) | 1 (1)
Hemorrage, GI-rectum (Gastrointestinal disorders) | 1 (1)
Pain-abdomen NOS (Vascular disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Cystitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neurgology-other: Delirium (altered mental status) (Psychiatric disorders) | 1 (1)
Other: Panhypopituitarism (Endocrine disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipilimumab and Androgen Depravation (N=27)
Abdominal Pain (Nervous system disorders) | 1 (2)
Adrenal Insufficiency (Renal and urinary disorders) | 1 (1)
Alanine Aminotransferase increased (Hepatobiliary disorders) | 1 (2)
Albumin, serum-low (hypoalbuminemia) (Hepatobiliary disorders) | 6 (8)
Alkaline phosphatase (Hepatobiliary disorders) | 13 (19)
Alkaline phosphatase increased (Hepatobiliary disorders) | 1 (1)
Allergy/Immunology-Other (Specify) (General disorders) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 16 (38)
Amylase (Gastrointestinal disorders) | 8 (12)
Anemia (Blood and lymphatic system disorders) | 3 (7)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (non-specific) (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 1 (1)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 16 (37)
Auditory/Ear-Other (Specify) (Ear and labyrinth disorders) | 1 (1)
Back pain (Nervous system disorders) | 3 (3)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 9 (12)
Bilirubin (hyperbilirubinemia) (Hepatobiliary disorders) | 5 (16)
Blood/Bone Marrow-Other (Specify) (Blood and lymphatic system disorders) | 10 (17)
Blurred vision (Eye disorders) | 1 (1)
Bone pain (Nervous system disorders) | 1 (1)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 2 (2)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 3 (3)
Cholesterol, serum-high (hypercholestremia) (Metabolism and nutrition disorders) | 1 (1)
CNS cerebrovascular ischemia (Vascular disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
Constitutional Symptoms-Other (Specify) (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Creatinine (Renal and urinary disorders) | 5 (9)
Cushingoid appearance (e.g., moon face, buffalo hump, centripetal obesity, cutaneous striae) (Endocrine disorders) | 1 (1)
Cystitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dermatology/Skin-Other (Specify) (Skin and subcutaneous tissue disorders) | 6 (10)
Diarrhea (Gastrointestinal disorders) | 14 (28)
Distension/bloating, abdominal (Gastrointestinal disorders) | 2 (4)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Gastrointestinal disorders) | 1 (1)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Edema: head and neck (Vascular disorders) | 3 (3)
Edema: limb (Vascular disorders) | 3 (17)
Endocrine-Other (Specify) (Endocrine disorders) | 4 (7)
Erectile dysfunction (Reproductive system and breast disorders) | 3 (3)
Fatigue (asthenia, lethargy, malaise) (Metabolism and nutrition disorders) | 22 (44)
Febrile neutropenia (Infections and infestations) | 1 (1) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10^9 per liter
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10^9 per liter) (Infections and infestations) | 4 (4)
Flank pain (Nervous system disorders) | 1 (1)
Flatulence (Musculoskeletal and connective tissue disorders) | 1 (2)
Flu-like syndrome (Infections and infestations) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal-Other (Specity) (Gastrointestinal disorders) | 3 (3)
GGT (gamma-Glutamyl transpeptidase) (Hepatobiliary disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 21 (56)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1)
Hair loss/alopecia (scalp or body) (Endocrine disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Hemoglobin (Blood and lymphatic system disorders) | 25 (56)
Hemoglobinuria (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage, GI--Select (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GU--Select (Kidney) (Renal and urinary disorders) | 1 (1)
Hot flashes (Endocrine disorders) | 1 (1)
Hot flashes/flushes (Endocrine disorders) | 15 (18)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Hypertension (Adult) (Cardiac disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Cardiac disorders) | 2 (3)
Incontinence, urinary (Renal and urinary disorders) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils--Select (Sinus) (Infections and infestations) | 1 (1)
Infection with unknown ANC--Select (Infections and infestations) | 1 (2)
Infection-Other (Specify) (Infections and infestations) | 4 (5)
Insomnia (Nervous system disorders) | 6 (11)
Investigations - Other, specify (Blood and lymphatic system disorders) | 1 (7)
Joint-function (Musculoskeletal and connective tissue disorders) | 2 (4)
Leukocytes (Total WBC) (Blood and lymphatic system disorders) | 6 (12)
Lipase (Metabolism and nutrition disorders) | 9 (18)
Localized edema (Vascular disorders) | 1 (1)
Lymphopenia (Vascular disorders) | 6 (9)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 9 (13)
Metabolic/Laboratory-Other (Specify) (Metabolism and nutrition disorders) | 2 (4)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Mood alteration--Select (Psychiatric disorders) | 1 (1)
Mood alteration--Select (Anxiety) (Psychiatric disorders) | 2 (2)
Mucositis/stomatitis (clinical exam) (Oral Cavity) (Gastrointestinal disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 4 (5)
Muscle weakness, generalized or specific area (not due to neuropathy) (Extremity - lower) (Musculoskeletal and connective tissue disorders) | 2 (4)
Muscle weakness, generalized or specific area (not due to neuropathy) (Whole body/generalized) (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal/Soft Tissue-Other (Specify) (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (7)
Nausea (Gastrointestinal disorders) | 9 (17)
Neurology-Other (Specify) (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Musculoskeletal and connective tissue disorders) | 6 (7)
Neutrophil count decreased (Metabolism and nutrition disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Metabolism and nutrition disorders) | 1 (5)
Ocular/Visual-Other (Specify) (Eye disorders) | 1 (1)
Pain (Nervous system disorders) | 3 (12)
Pain-Other (Specify) (Nervous system disorders) | 14 (34)
Pain--Select (Nervous system disorders) | 2 (2)
Pain--Select (Abdomen NOS) (Nervous system disorders) | 1 (1)
Pain--Select (Back) (Nervous system disorders) | 5 (5)
Pain--Select (Extremity-limb) (Nervous system disorders) | 1 (3)
Pain--Select (Head/headache) (Nervous system disorders) | 4 (8)
Pain--Select (Joint) (Nervous system disorders) | 1 (2)
Pain--Select (Kidney) (Nervous system disorders) | 1 (1)
Pain--Select (Pain NOS) (Nervous system disorders) | 1 (1)
Pain--Select (Pelvis) (Nervous system disorders) | 2 (2)
Pain--Select (Prostate) (Nervous system disorders) | 1 (1)
Pain--Select (Rectum) (Nervous system disorders) | 2 (2)
Paresthesia (Skin and subcutaneous tissue disorders) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (2)
Platelets (Respiratory, thoracic and mediastinal disorders) | 5 (11)
Pneumonitis/pulmonary infiltrates (Metabolism and nutrition disorders) | 1 (1)
Potassium serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (3)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3 (5)
Proteinuria (Metabolism and nutrition disorders) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1)
Pulmonary/Upper Respiratory-Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 18 (40)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (2)
Renal/Genitourinary-Other (Specify) (Renal and urinary disorders) | 3 (3)
Rigors/chills (Nervous system disorders) | 1 (1)
Sodium serum-low (hyponatremia) (Metabolism and nutrition disorders) | 8 (11)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 2 (2)
Supraventricular and nodal arrhythmia--Select (Sinus bradycardia) (Cardiac disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Thyroid function, high (hyperthyroidism, thyrotoxicosis) (Endocrine disorders) | 4 (4)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 10 (12)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 16 (18)
Vision-blurred vision (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (9)
Watery eye (epiphora, tearing) (Eye disorders) | 3 (3)
Weight gain (Metabolism and nutrition disorders) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 3 (4)
White blood cell decreased (Blood and lymphatic system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-02-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT01377389/Prot_SAP_000.pdf